CLINICAL TRIAL: NCT00610883
Title: LSA4 Protocol for the Treatment of Advanced Pediatric and Adolescent Non-Hodgkins Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90-042
Record Dates: First submitted 2007-12-26; First posted 2008-02-08 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Cyclophosphamide; Methotrexate; Daunorubicin; Asparaginase; Carmustine

ARMS (1):
- 1 - LSA4 (Experimental)
  Interventions: Drug: LSA4, Cyclophosphamide, Methotrexate, Daunomycin, L-asparaginase, BCNU

INTERVENTIONS:
Drug: LSA4, Cyclophosphamide, Methotrexate, Daunomycin, L-asparaginase, BCNU — LSA4 intervention includes three phases: induction, consolidation and maintenance

SUMMARY:
Non-Hodgin's lymphoma is curable in 76% of patients. In nonlymphoblastic lymphmas, cancer may return on average 3 months from beginning treatment and for lymphoblastic lymphomas, 6 months. To aggressively treat this cancer this study uses effective drugs in three parts:

* Induction ends on day 19
* Consolidation ends on day 38 or 42
* Maintenance may include up to 6 cycles

ELIGIBILITY:
Inclusion Criteria:

* Non-Hodgkin's Lymphoma stages III, IV, IVA with

  1. T cell lymphomas, any primary site irrespective of LDH level
  2. large cell lymphomas, any primary site irrespective of LDH level
  3. B cell lymphomas, any primary site with initial LDH of less than 500

Exclusion Criteria:

* B cell lymphomas, any primary site with initial LDH of less than 500 and initial CNS or bone involvement

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 1990-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Trippett, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: LSA4, Cyclophosphamide, Methotrexate, Daunomycin, L-asparaginase, BCNU: LSA4 intervention includes three phases: induction, consolidation and maintenance
Period: Overall Study
Arm/Group | All Patients
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 17
Age, Customized [Median (Full Range); unit: years]
  Median Age | 12 [2 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission
Description: The number of patients who achieved a complete remission as a result of treatment
Time Frame: 330 Days
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 17
participants | 10

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=17)
Ruptured Necrotic Tumor (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=17)
Hematological Toxicity (Blood and lymphatic system disorders) | 17 (17)
Hepatic Toxicity (Renal and urinary disorders) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes